CLINICAL TRIAL: NCT04715061
Title: Modulation of Immune Response and Side Effects of Cancer Treatments by Aerobic Exercise: Role of Exercise Intensity
Brief Title: Impact of Aerobic Exercise on Immune Response and Side Effects of Cancer Treatments
Acronym: CANEX-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-3547
Record Dates: First submitted 2020-12-11; First posted 2021-01-20 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer Stage IV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Each participant performed 3 experimental conditions (rest, moderate continuous training and interval training).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cancer patients with MRI (Experimental): 9 cancer patients will be recruited and received the 3 experimental conditions : first the rest condition (with MRI), then randomly MICE condition and HIIT condition (with MRI).
  Interventions: Other: Resting state (Control); Other: Moderate Intensity Continuous Exercise (MICE); Other: High Intensity Interval Exercise (HIIE)
- Cancer patients without MRI (Experimental): 9 cancer patients will be recruited and received the 3 experimental conditions : first the rest condition, then randomly MICE condition and HIIT condition, all without MRI.
  Interventions: Other: Resting state (Control); Other: Moderate Intensity Continuous Exercise (MICE); Other: High Intensity Interval Exercise (HIIE)
- Healthy patients (Active Comparator): 9 healthy patients will be recruited and received 2 experimental conditions : first the rest condition (with a MRI), then HIIT condition (with MRI).
  Interventions: Other: Resting state (Control); Other: High Intensity Interval Exercise (HIIE)

INTERVENTIONS:
Other: Resting state (Control) — Participants were asking to sit on a sofa for 50 minutes.
Other: Moderate Intensity Continuous Exercise (MICE) — MICE condition consisted of 50 minutes of moderate and continuous aerobic exercise on ergocycle. This includes a warm-up and cool-down period at low intensity, and a 40-minute period at moderate intensity (power output is equivalent to an effort perception from 4 to 6/10 and lactate levels from 2 to 4 mmol/L, obtained by submaximal test)
  Arms: Cancer patients with MRI; Cancer patients without MRI
Other: High Intensity Interval Exercise (HIIE) — HIIT condition consisted of a 30 minutes of aerobic exercise training perform on ergocycle. This includes a warm-up at low intensity, followed by 10 blocks of 1 minute at high intensity (power output corresponding to the highest power reached at the submaximal test and lactate levels > 4 mmol/L) and 1 minute of active cooldown (effort perception around 1-2/10).

SUMMARY:
Aerobic exercise is associated with many benefits in patients with cancer treatments. Among these, the reduction of cancer-related fatigue (CRF) is one of the best demonstrated. Besides, several animal models have shown a marked reduction in tumor growth with aerobic exercise, sometimes by more than 60%. As the level of physical activity is convincingly associated with a reduction in the risk of cancer or recurrences, this suggests that aerobic exercise may represent a central therapeutic approach during treatment, both against CRF and for its potential anti-tumor effect.

Both benefits have been suggested to be based on the immunostimulatory and anti-inflammatory effects of exercise. Indeed, systemic inflammatory activity seems to play a central role in the etiology of CRF during cancer treatments, among other things by stimulating the neuro-inflammatory activity of the central nervous system. Also, regarding the anti-tumor effect of exercise, animal models show that this benefit is partly explained by an increase in the activity of immune cells called natural killers (Natural Killer; NK) in tumor tissue and a reduction in the activity of regulatory T cells, the latter having an immunosuppressive effect. However, in humans, the results vary. While some improvement in NK cell activity has been reported in response to aerobic training in breast cancer survivors, others have seen no effect on the immune profile of patients and survivors. On the other hand, some authors report an improvement in the inflammatory profile with training, while others report little or no effect, as well as weak associations with the perception of fatigue.

Although these results seem to discredit the hypothesis of immune and inflammatory regulation of exercise in humans, these studies have all looked at the effect of several weeks of training on the inflammatory and immune profile on an empty stomach and rest. However, several results from the field of exercise immunology convincingly show that the anti-inflammatory effect, as well as the immunostimulating effect of aerobic exercise (including the anti-tumor activity of NK cells) are mainly acute and transient, ie. in the hours following the end of the effort. Furthermore, certain results suggest that in the context of chemotherapy treatments, cyclical treatment by nature, the peaks of fatigue are also acute (i.e. in the days following the treatment) and parallel to peaks of inflammatory activity.

Considering these results, it is therefore plausible to assume that the effect of aerobic exercise on suppressing tumor growth and reducing CRF results rather than the repetition of this acute response at each exercise session. In this case, the prescription of aerobic exercise preceding a session of chemotherapy could potentially represent an interesting therapeutic modality, allowing both the reduction of the CRF associated with this treatment, as well as a better response to the treatment. Besides, as this acute response seems to be highly dependent on the intensity of the effort, high-intensity interval training (HIIT) could be a particularly interesting approach in this context, because it does not require that the high intensity or long-lasting exercise. However, considering the immunosuppressive and pro-inflammatory effects of chemotherapy, the extent of the acute response to exercise may not allow this type of therapeutic use to be considered in this population. To date, no study has attempted to characterize the acute immune and inflammatory response following aerobic exercise in patients currently undergoing chemotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic colorectal cancer
* At the beginning of their chemotherapy treatment
* Eastern Cooperative Oncology Group (ECOG) performance status between grades 0 to 1
* Physically capable to realise HIIT and continous moderate aerobic exercise on ergocycle

Exclusion Criteria:

* Orthopedic, cardiac or metabolic limitations preventing aerobic effort
* Betablockers
* Surgery planned for the next two months following recruitment

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Change in the concentration of different peripheral blood mononuclear cells (Natural Killer Cells, T cells and monocytes) | Before the start of the condition (t = 0 minute), at the end of the condition (t = 50 minutes), 1 hour post-condition (t = 110 minutes)
  Flow cytometry

SECONDARY OUTCOMES:
Change in the concentration of inflammatory mediators in peripheral blood (chemokines, pro- and anti-inflammatory cytokines) | Before the start of the condition (t = 0 minute), At the end of the condition (t = 50 minutes), 1 hour post-condition (t = 110 minutes), 2 hour post-condition (t = 170 minutes)
  Luminex immunoassay
Change of hormonal profile (cortisol, corticotropin-releasing hormone (CRH), adrenocorticotropic hormone (ACTH), adrenaline and noradrenaline) | Before the start of the condition (t = 0 minute), At the end of the condition (t = 50 minutes), 1 hour post-condition (t = 110 minutes), 2 hour post-condition (t = 170 minutes)
  ELISA Kits and Salivary Cortisol Enzyme ImmunoAssay Kit
Change of Indoleamine-2,3-Dioxygenase activation | Before the start of the condition (t = 0 minute), At the end of the condition (t = 50 minutes), 1 hour post-condition (t = 110 minutes), 2 hour post-condition (t = 170 minutes)
  Liquid chromatography-mass spectrometry (LCMS)
Cancer-Related Fatigue | During 5 days after the day of the condition, 3 times per day
  Visual Analogue Scale, graduated from 0 (no fatigue) to 10 (extreme fatigue)
Cerebral integrity - Cerebral blood flow | At the end of the condition (t = 50 minutes) within a 30-minute time window
  Functional MRI (pcASL technique)
Heart rate variability | At the end of the condition, during 10 minutes (t = 50 minutes to t = 60 minutes)
  Heart rate monitor

CONTACTS AND LOCATIONS:
Locations (1):
- Research Centre on Aging, Sherbrooke, Quebec, Canada